CLINICAL TRIAL: NCT06043115
Title: Factors Affecting Mortality in Covid-19 Disease
Status: Completed | Type: Observational
Sponsor: Melike Cengiz (Other)
Responsible Party: Sponsor-Investigator, Melike Cengiz, MD,Professor Doctor, Akdeniz University
Organization: Akdeniz University (Other)
Other Study IDs: Akdeniz University Faculty
Record Dates: First submitted 2023-09-09; First posted 2023-09-21 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: COVID-19 Pneumonia; Mortality

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- covid-19 survival cohort: consists of surviving patients
  Interventions: Other: covid-19 survival cohort
- covid-19 mortality cohort: consists of deceased patients
  Interventions: Other: covid-19 mortality cohort

INTERVENTIONS:
Other: covid-19 survival cohort — consists of surviving patients
  Groups: covid-19 survival cohort
Other: covid-19 mortality cohort — consists of deceased patients
  Groups: covid-19 mortality cohort

SUMMARY:
The coronavirus disease-19 (COVID-19), defined by the reporting of pneumonia cases of unknown etiology at the end of 2019 in Wuhan, China, has spread worldwide, causing millions of deaths. Despite the fact that more than two years have passed since the struggle against the disease it continues to be an important public health problem.The increasing number of critically ill patients with this pandemic caused a great demand for intensive care units (ICU), and ICU capacity and staff had to be rapidly expanded in many countries. Similarly, in various periods of the pandemic in Turkey, the capacity of many ICUs had to be increased. The rates of admission to the ICU and death rates differed greatly from center to center due to various factors such as ICU bed capacity and the duration of access to the ICU, patient characteristics, and differences in the treatments applied. Determining the factors that may be associated with mortality is important in terms of improving the ICU follow-up of patients with COVID-19 and guiding their treatment.There is limited information about the characteristics and mortality of Turkish patients with COVID-19 in the ICU. The aim of this study is to determine the demographic, clinical and laboratory characteristics and the factors affecting ICU mortality in COVID-19 patients followed in Akdeniz University Medical Faculty Hospital since the beginning of the pandemic.

DETAILED DESCRIPTION:
It was designed as a retrospective cohort study in which patients with a diagnosis of COVID-19 hospitalized in the ICU between 11 March 2020 and 31 March 2022 were included.

Patients aged ≥18 years with a confrmed diagnosis of the severe acute respiratory syndrome coronavirus-2 (SARS-CoV-2) infection by a positive real-time reverse-transcription polymerase chain reaction test (RT-PCR) on a nasopharyngeal swab or or endotracheal aspirate were included in the present study. The study data collected from the patient record at ICU admission included demographic characteristics (age, sex, body mass index), smoking history, comorbidities, vaccination status, Acute Physiology and Chronic Health Evaluation II (APACHE II) score, Sequential Organ Failure Assessment (SOFA) score, laboratory findings, blood gas analysis (PaO2/FiO2 ratio), oxygen device method, lenght of stay ICU and hospital duration and COVID-19 related complications. Laboratory findings included a complete blood count, coagulation testing, D-dimer, blood chemical analysis, C-reactive protein (CRP), assessment of liver and renal function, procalcitonin, and microbial cultures results. Additional adjunctive support, including extracorporeal membrane oxygenation (ECMO), prone positioning, renal replacement therapy (RRT) were documented daily. Information on patient-specific therapies, such as administration of hydroxychloroquine, antivirals, convalescent plasma and plasmapheresis was also collected.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥18 years with a confrmed diagnosis of the severe acute respiratory syndrome coronavirus-2 infection by a positive real-time reverse-transcription polymerase chain reaction test

Exclusion Criteria:

* Patients whose SARS-CoV-2 RT-PCR test was negative
* Chest computed tomography findings or symptoms were not compatible with COVID-19

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged ≥18 years with a confrmed diagnosis of the severe acute respiratory syndrome coronavirus-2 (SARS-CoV-2) infection by a positive real-time reverse-transcription polymerase chain reaction test (RT-PCR) on a nasopharyngeal swab or endotracheal aspirate were included in the present study.
Sampling Method: Non-Probability Sample
Enrollment: 619 (Actual)
Dates: Start 2022-05-11 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2022-12-15 (Actual)

PRIMARY OUTCOMES:
factors affecting mortality in COVID-19 | 11 March 2020 -31 March 2022
  clinical and laboratory characteristics of COVID-19 patients in mortality of ICU.

SECONDARY OUTCOMES:
difference between the pandemic waves | 11 March 2020-31 March 2022
  mortality rate of ICU, clinical and laboratory characteristics of COVID-19 patients according to pandemic waves

CONTACTS AND LOCATIONS:
Overall Officials: Burcu Ozer, MD, Principal Investigator — Akdeniz University School of Medicine, Department of Anesthesiology and Reanimation, Turkey
Locations (1):
- Akdeniz University School of Medicine, Department of Anesthesiology and Intensive Care, Turkey, Antalya, Turkey (Türkiye)